CLINICAL TRIAL: NCT05535868
Title: Serotype 3 Experimental Human Pneumococcal Challenge; Dose Ranging and Reproducibility in a Healthy Volunteer Population
Brief Title: Experimental Human Pneumococcal Challenge With SPN3
Acronym: Challenge3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-003
Record Dates: First submitted 2022-04-14; First posted 2022-09-10 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Streptococcus Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPN3. (Experimental): Inoculation with SPN3 at D0 visit. 0.1ml of pneumococcus is given
  Interventions: Other: SPN3 innoculation
- SPN3 booster (Experimental): inoculation booster at day 14 This visit will only occur for participants who have tested negative for SPN3 at days 2 and 7. 0.1ml of pneumococcus is given
  Interventions: Other: SPN3 innoculation

INTERVENTIONS:
Other: SPN3 innoculation — Healthy adult participants aged 18-50 (inclusive) will be inoculated with pure culture of well-characterised, fully sequenced amoxicillin-sensitive SPN3. They will be observed for safety and development of pneumococcal colonisation

SUMMARY:
The 'Experimental Human Pneumococcal challenge' (EHPC) model is a way of putting drops of bacteria into the nose. Investigators have studied this model of putting bacteria in the nose safely in over 1500 volunteers over the past decade with no serious side effects and now want to test the model using a different strain of the bacteria that is commonly found in the community, SPN3.

The aim of this study is to determine how much pneumococcus is needed to achieve nasal colonisation and how long the bacteria live in the nose for before natural immune responses eradicate them. By doing this, Investigators will then be able to test how well future vaccines prevent colonisation with pneumococcus. Investigators want to learn more about how the immune system responds to nasal colonisation with pneumococcus, again to help with development of new vaccines.

DETAILED DESCRIPTION:
In this study, investigators propose to determine the optimal dose and isolate of SPN3 to establish colonisation in the human nasopharynx, as well as improving knowledge of immune responses to SPN3 colonisation. The results from this study will be used to inform development of improved SPN3 vaccines and to inform design of future pneumococcal vaccine RCTs.

To increase the relevance of the EHPC model and its use for assessing future vaccines such as V114, investigators are proposing here to set up an EHPC model with carefully selected non-proprietary SPN3 strains. Investigators will conduct a safety and dose-ranging study to determine the optimum SPN3 strain and dose for colonisation acquisition and confirm the dose in a subsequent larger cohort in a reproducibility study and will study mucosal and systemic immune responses to this serotype and their association with protection against colonisation acquisition and clearance.

ELIGIBILITY:
Inclusion Criteria:• Healthy young adults aged 18-50 years (inclusive). This age range minimises the risk of invasive pneumococcal infection and allows comparison with previously published experimental work done by our group.

* Fluent spoken English - to ensure a comprehensive understanding of the research project and their proposed involvement, enabling valid consent to be given.
* Access to their own mobile telephone - to ensure safety and timely communication.
* Capacity to give informed consent.

Exclusion Criteria:

* o Currently involved in another study unless observational or non-interventional, excluding the EHPC bronchoscopy study (at the discretion of the study team). This is to ensure no harm comes to the participants through over-sampling.

  * Participant in any previous EHPC trial in past year
  * Participant in previous EHPC trial inoculated with SPN3 in the last 3 years
  * Participant in EHPC Pneumo 2 trial

    * Vaccination: Previous pneumococcal vaccination PPV23 or PCV13 (routine in babies born in the UK since 2005) or PCV10. This can be self-reported or confirmed from GP questionnaire (GPQ) if deemed necessary at clinician discretion.
    * Allergy: to penicillin/amoxicillin
    * Health history (self-reported or confirmed by GPQ or medical summary if felt to be necessary at clinician discretion):
  * Chronic ill health including immunosuppressive history, diabetes, asthma (on regular medication), recurrent otitis media or other respiratory disease.
  * Medication that may affect the immune system e.g., steroids, inflammation altering or disease-modifying anti-rheumatoid drugs.
  * Long term use of antibiotics for chronic infection.
  * Major pneumococcal illness requiring hospitalisation in the last 10 years.
  * Other conditions considered by the clinical team as a concern for participant safety or integrity of the study
  * Significant mental health problems (uncontrolled condition or requiring previous admission to a psychiatric unit) that would impair ability to participate

    • Direct caring role or close contact with individuals at higher risk of infection during the inoculation period if personal protective equipment (PPE) not worn:
  * Children under 5 years age
  * Adults with chronic ill health or immunosuppression
  * Hospital patients

    • Smoker:
  * Current or ex-smoker (daily cigarettes, daily e-cigarettes/vaping and daily smoking of recreational drugs) in the last 6 months. Participants who smoke <5 cigarettes per week may be included.
  * Previous significant smoking history (>20 cigarettes per day for 20 years or equivalent [>20 pack years]).

    • Biologically female participants of child-bearing potential (WOCBP) who are:
  * Currently pregnant/lactating
  * Intending on becoming pregnant during the study
  * Not deemed to have effective birth control

    • History of or current drug or alcohol abuse:
  * Men should not drink >3 units/day regularly
  * Women should not drink >2 units/day regularly

    * Overseas travel planned in follow up period of study visits
    * Natural SPN 3 colonisation in baseline nasal wash - if a participant is colonised with non-SPN3 pneumococcus, they can be included as part of exploratory analyses, but would not be included in the primary analysis
    * STOP criteria - participants who meet STOP criteria at time of screening (Table 3) 6.3 Temporary Exclusion Criteria
    * Ongoing COVID-19 symptoms (fever, cough, shortness of breath, anosmia or ageusia) or confirmed current COVID-19 infection. Participants with resolved COVID-19 after their UKHSA determined isolation period has ended can be included.
    * Current/acute illness within 14 days prior to inoculation if COVID-19 negative
    * Positive COVID-19 swab whether symptomatic or asymptomatic within 10 days of inoculation
    * Currently isolating following exposure to COVID-19 as per UKHSA guidance
    * Antibiotic use within 28 days of inoculation.
    * Participants who have been temporarily excluded at screening may be re-screened at a later date to assess their eligibility at this time for inclusion into the study. At this point, the participant would be re-consented if their initial written consent was given >4 months prior to this date.
    * Vaccination 21 days prior to inoculation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with experimental SPN3 colonisation of the nasopharynx (assessing change from non carrier to carrier) | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 2,7,13,16,21 or day 28
  change from non carrier to carrier determined by SPN3 presence in classical microbiological culture in at least one nasal wash (NW) sample, at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.

SECONDARY OUTCOMES:
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individually atday 0 or day 14 or both)) ie day 2,
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 7
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individuallyat day 0 or day 14 or both) ) ie day 13
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 16
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 21
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The rate of occurrence of SPN3 experimental colonisation of the nasopharynx | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both) ) ie day 28
  determined by SPN3 presence in classical microbiological culture and qPCR (combined and individually) from at least one NW sample at any time point following one or two inoculations (combined and individually). This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 2
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day ,7,
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both) ) ie day 13
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both)) ie day 16
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both) ) ie day 21
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The bacterial density of experimental SPN3 colonisation of the nasopharynx in NW, at each and any time point following one or two inoculations (combined and individually), | at any time point following one or two inoculations (combined and individually at day 0 or day 14 or both) ) ie day 28
  determined by classical microbiological culture and molecular methods. This will be assessed for each isolate and dose separately.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually at day 0 or day 14 or both)) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 2
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 7
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually at day 0 or day 14 or both)) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 13
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually at day 0 or day 14 or both)) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 16
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually at day 0 or day 14 or both)) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 21
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.
The duration of experimental SPN3 colonisation of nasopharynx | The timepoint last NW sample following one or two inoculations (combined and individually at day 0 or day 14 or both)) in which SPN3 is detected by classical microbiological culture or molecular methods ie day 28
  determined by the last NW sample following one or two inoculations (combined and individually) in which SPN3 is detected by classical microbiological culture or molecular methods.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Collins, MBChB, PhD, Principal Investigator — Senior Clinical Lecturer
Locations (1):
- LSTM, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No